CLINICAL TRIAL: NCT02227017
Title: An Open-label, Single-site, One-sequence Cross-over Study to Assess the Relative Bioavailability of TPV/r 500 mg/200 mg at Steady State When TPV and RTV Are Administered as Oral Solutions vs. Capsules in the Fed and Fasted State.
Brief Title: Relative Bioavailability of Tipranavir (TPV)/Ritonavir (RTV) at Steady State Administered as Oral Solutions vs. Capsules in the Fed and Fasted State in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1182.100
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Ritonavir

ARMS (4):
- TPV/RTV capsules fed (Experimental)
  Interventions: Drug: TPV capsule; Drug: RTV capsule; Other: standard meal
- TPV/RTV capsules fasted (Experimental)
  Interventions: Drug: TPV capsule; Drug: RTV capsule
- TPV/RTV solutions fed (Active Comparator)
  Interventions: Drug: TPV solution; Drug: RTV solution; Other: standard meal
- TPV/RTV solutions fasted (Active Comparator)
  Interventions: Drug: TPV solution; Drug: RTV solution

INTERVENTIONS:
Drug: TPV capsule
  Arms: TPV/RTV capsules fasted; TPV/RTV capsules fed
Drug: TPV solution
  Arms: TPV/RTV solutions fasted; TPV/RTV solutions fed
Drug: RTV capsule
  Arms: TPV/RTV capsules fasted; TPV/RTV capsules fed
Drug: RTV solution
  Arms: TPV/RTV solutions fasted; TPV/RTV solutions fed
Other: standard meal
  Arms: TPV/RTV capsules fed; TPV/RTV solutions fed

SUMMARY:
Study to establish the relative bioavailability of the TPV oral solution formulation (500 mg coadministered with RTV oral solution 200 mg) to the TPV capsule formulation (500 mg coadministered with RTV capsules 200 mg), with both treatments at steady-state under fasted and fed conditions in healthy male and female volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 to 65 years of age inclusive
2. A Body Mass Index (BMI): ≥18.5 and ≤35 kg/m2
3. Signed informed consent prior to performance of any study procedures
4. Ability to swallow multiple large capsules without difficulty
5. Screening laboratory values within the normal range. Inclusion of any subject with an abnormal laboratory value was subject to approval by the BI trial clinical monitor
6. Acceptable medical history, physical examination, and 12-lead ECG at screening
7. Willingness to abstain from the following starting 5 days prior to administration of any study medication and up until the end of the study:

   * Grapefruit or grapefruit juice, red wine, Seville oranges, St. John's Wort and Milk Thistle
8. Willingness to abstain from the following starting 3 days prior to administration of any study medication up to the end of the study:

   * Garlic supplements and methylxanthine containing foods or drinks (including coffee, tea, cola, energy drinks, chocolate, etc.), apples and apple juice
9. Willingness to abstain from over-the-counter herbal medications for the duration of the study
10. Are non-smokers
11. Willingness to abstain from vigorous physical exercise during intensive pharmacokinetic days 10, 11, 14, 15
12. Reasonable probability for completion of the study

Exclusion Criteria:

1. Participation in another trial with an investigational medicine within 2 months prior to Day 0 of this study
2. Female subjects of reproductive potential who:

   * Have a positive pregnancy test
   * Have not been using a barrier method of contraception for at least 3 months prior to participation in the study
   * Are not willing to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and 60 days after completion/termination of the trial
   * Are breast-feeding
   * Use any pharmacological contraceptive (including oral, patch or injectable contraceptives) within 1 month prior to Day 0 and for the duration of the study. Due to long half-life, subjects using Depo-Provera® within 6 months prior to Day 1 are excluded from participation in this study
   * Use of hormone replacement therapy within 1 month prior to Day 0 and anytime during the study
3. Use of any medication listed in Protocol within 30 days prior to Day 0 of this study
4. Administration of antibiotics within 15 days prior to Day 0 and anytime during the study
5. History of acute illness within 60 days prior to Day 0

   * Subjects will be excluded for acute illnesses that occurred more than 60 days prior to Day 0 if, in the opinion of the investigator, the subject did not qualify as a healthy volunteer
6. Serological evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV)
7. Serological evidence of exposure to HIV
8. Alcohol or substance abuse within 1 year prior to screening or during the study
9. Blood or plasma donations within 30 days prior to Day 0 or during the study
10. Subjects with a history of any illness or allergy that, in the opinion of the investigator, might have confounded the results of the study or pose additional risk in administering TPV, or RTV to the subject
11. Subjects who have taken (within 7 days prior to Day 0) any over-the-counter or prescription medication that, in the opinion of the investigator in consultation with the sponsor's clinical monitor, might have interfered with absorption, distribution, or metabolism of the study medications
12. Known hypersensitivity to sulphonamide class of drugs
13. Known hypersensitivity to TPV, RTV, or antiretroviral drugs (marketed or experimental use as part of clinical research studies)
14. Known elevated liver enzymes in past trials with any compound
15. Known allergy to nuts or nut products (A spoonful of peanut or hazelnut butter was taken immediately before administration of TPV or RTV oral solution, to help mask the taste of the solutions)
16. Inability to adhere to the protocol
17. Inability to consume a standard high-fat meal
18. Cautions or warnings in the package insert which, in the opinion of the investigator, constituted grounds for subject exclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-02; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of TPV from time zero to 12 hours at steady state (AUC0-12) | up to 12 hours after drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of RTV from time zero to 12 hours at steady state (AUC0-12) | up to 12 hours after drug administration
Maximum measured concentration of the analyte in plasma at steady state (Cmax) | up to 12 hours after drug administration
Drug concentration in plasma after 12 hours at steady state (Cp12h) | up to 12 hours after drug administration
  Drug concentration in plasma at last measurement (Cplast) if Cp12h is below limit of quantification (BLQ)
Apparent clearance of the analyte in plasma at steady state following extravascular administration (CL/F) | up to 12 hours after drug administration
Volume of distribution at steady state (Vd) | up to 12 hours after drug administration
Terminal half life at steady state (t1/2) | up to 12 hours after drug administration
Number of subjects with adverse events | up to day 16
Number of subjects with clinically significant findings in vital signs | up to day 16
  blood pressure, pulse rate
Number of subjects with clinically significant findings in ECG | up to day 16
Number of subjects with clinically significant findings in laboratory tests | up to day 16